CLINICAL TRIAL: NCT06840457
Title: COMPASS: Comprehensive Mobile Precision Approach for Scalable Solutions in Mental Health Treatment
Brief Title: COMPASS: a Comprehensive Mobile Precision Approach for Scalable Solutions in Mental Health Treatment
Acronym: COMPASS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Amy S.B. Bohnert, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00248932; 1U01MH136025 (NIH)
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Mental Health
MeSH Terms: conditions — Psychological Well-Being | interventions — Mindfulness; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Mindfulness with tailored messages (Active Comparator): Participants will receive an app-based intervention, tailored messages from the MyDataHelps study app, and activity tracker.
  Interventions: Behavioral: Mindfulness + Tailored Messages
- Mindfulness without tailored messages (Active Comparator): Participants will receive an app-based intervention and standard feedback from activity tracker.
  Interventions: Behavioral: Mindfulness without Tailored Messages
- Cognitive Behavioral Therapy (CBT) with tailored messages (Active Comparator): Participants will receive an app-based intervention, tailored messages from the MyDataHelps study app, and activity tracker.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT) + Tailored Messages
- Cognitive Behavioral Therapy (CBT) without tailored messages (Active Comparator): Participants will receive an app-based intervention and standard feedback from activity tracker.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT) without Tailored Messages

INTERVENTIONS:
Behavioral: Mindfulness + Tailored Messages — Tailored Messages (TM) Participants randomized to receive enhanced feedback will receive this feedback from the MyDataHelps study app. This includes varying types of text and visual feedback based on data collected through the app. Messages will be displayed to participants on a dashboard in the app or delivered via pop-up notifications. Participants will receive a combination of text and visual messages.
  The study will use an app designed to train the user in mindfulness practices.
  Other Names: Mindfulness
  Arms: Mindfulness with tailored messages
Behavioral: Mindfulness without Tailored Messages — The study will use an app designed to train the user in mindfulness practices.
  Other Names: Mindfulness
  Arms: Mindfulness without tailored messages
Behavioral: Cognitive Behavioral Therapy (CBT) + Tailored Messages — Tailored Messages (TM) Participants randomized to receive enhanced feedback will receive this feedback from the MyDataHelps study app. This includes varying types of text and visual feedback based on data collected through the app. Messages will be displayed to participants on a dashboard in the app or delivered via pop-up notifications. Participants will receive a combination of text and visual messages.
  The study will use an app designed to deliver cognitive behavioral therapy.
  Other Names: CBT
  Arms: Cognitive Behavioral Therapy (CBT) with tailored messages
Behavioral: Cognitive Behavioral Therapy (CBT) without Tailored Messages — The study will use an app designed to deliver cognitive behavioral therapy.
  Other Names: CBT
  Arms: Cognitive Behavioral Therapy (CBT) without tailored messages

SUMMARY:
This research study is being conducted to understand if patients benefit from mobile health interventions while waiting for in-clinic mental health treatments.

ELIGIBILITY:
Inclusion Criteria:

* Seeking mental health services from Michigan Medicine, University Health Services, or collaborative clinics and services.
* Must have daily access to a smartphone version that is compatible with study activity trackers.
* Understands English to enable consent and use of the MyDataHelps app and app-based interventions

Exclusion Criteria:

* Self-reported or medical record indication of a current eating disorder
* Unable to provide informed consent (e.g., cognitive or guardianship restrictions)
* Scheduled outpatient mental health appointment is a pediatric appointment (even if age 18+)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4400 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Depression as measured by the Patient Health Questionnaire 9(PHQ-9) | From enrollment to the 6-week assessment.
  The PHQ-9 is an instrument for screening, diagnosing, monitoring and measuring the severity of depression: The PHQ-9 incorporates self-report questions on 9 specific depression symptoms that align with the DSM-IV depression diagnostic criteria. PHQ-9 scores range from 0-27 and 27 indicates severe depression.
Anxiety as measured using the Generalized Anxiety Disorder 7-Item (GAD-7) Scale | From enrollment to the 6-week assessment.
  GAD-7 consists total score for the seven items ranges from 0 to 21. Scores of 5, 10, and 15 represent cut points for mild, moderate, and severe anxiety, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Shared within National Institute of Mental Health Data Archive via grant data collaborator core.